CLINICAL TRIAL: NCT01184287
Title: A Phase II Trial of Addition of Ranpirnase(ONCONASE®) to Permetrexed Plus Carboplatin in Patientes With Non-Squamous Non-Small Cell Lung Cancer
Brief Title: A Study Of Ranpirnase(Onconase®) To Pemetrexed Plus Carboplatin In Patients With Non-Squamous Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Program discontinued
Sponsor: Tamir Biotechnology, Inc. (Industry)
Responsible Party: Charles Muniz, Tamir Biotechnology, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P30-800
Record Dates: First submitted 2010-08-17; First posted 2010-08-18 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer, NSCLC, Lung Cancer; Previously untreated Non-Squamous, Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — ranpirnase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ranpirnase (Experimental): All patients who do not progress after two cycles of pemetrexed-carboplatin will receive the study drug, ranpirnase
  Interventions: Drug: Ranpirnase

INTERVENTIONS:
Drug: Ranpirnase — Cycles 3 and until patient progression, on days 1,8 and 15 in a 21 day cycle
  Other Names: Onconase

SUMMARY:
The purpose of the trial is to determine the rate of improvement in objective tumor response, following the addition of ranpirnase to ongoing pemetrexed-carboplatin chemotherapy, for patients with SD or PR following 2 cycles of doublet chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* ECOG less than 2
* Estimated survival of greater than 12 weeks

Exclusion Criteria:

* Prior systemic chemotherapy for locally advanced or metastatic NSCLC
* Use of any investigational agent within 28 days prior to registration
* Known hypersensitivity to any of the study drugs
* Brain metastases or leptomeningeal disease
* History of prior malignancy within the past three years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Response | 4 or more months
  To determine the rate of improvement in objective tumor response, following the addition of ranpirnase to ongoing pemetrexed-carboplatin chemotherapy, for patients with SD or PR following 2 cycles of doublet chemotherapy

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 2 years
  To determine the PFS in patients with SD, PR or CR following 2 cycles of doublet chemotherapy
Survival | 2 years
  To determine the survival of patients with SD, PR or CR following 2 cycles of doublet chemotherapy

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Van Andel Research Institute, Grand Rapids, Michigan
  - Sletten Cancer Specialists, Great Falls, Montana
  - The Cancer Institute at NYU Langone Medical Center, New York, New York
  - Tri-county Hematology-Oncology Associates, Inc, Canton, Ohio
  - Northern Utah Associates, Ogden, Utah